CLINICAL TRIAL: NCT06451263
Title: Nudge to Referral of Adnexal Masses to Gynecologic Oncology
Brief Title: Nudge to Gynecologic Oncology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Anna Jo Bodurtha Smith, MD, MPH, MSc, Gynecologic Oncology Instructor, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 27823; 854677 (Other: University of Pennsylvania)
Record Dates: First submitted 2024-05-31; First posted 2024-06-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: abnormal adnexal mass
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nudge (Experimental): The study consists of one intervention, a clinician nudge to gynecologic oncology referral.
  Interventions: Behavioral: Nudge

INTERVENTIONS:
Behavioral: Nudge — Referral to gynecologic oncology is recommended when patients are diagnosed with a complex adnexal mass on imaging (i.e., O-RADS 4 or 5 on ultrasound or MRI, Codex 4 or 5 on CT). When patients are identified as having an adnexal mass, the order will be pended by the clinical research coordinator and sent to the ordering provider with a message to sign. The order will be pended within 48 hours of resulting imaging. The message will include content about national guidelines on referral to gynecologic oncology with opt-out framed language.

SUMMARY:
Ovarian cancer lacks an effective screening test, and prompt treatment at diagnosis is the only way to improve outcomes. Referral to gynecologic oncology at diagnosis of adnexal mass is recommend by guidelines from every major medical organization. Yet, 1 in 4 patients with ovarian cancer nationwide and at Penn Medicine never see a gynecologic oncologist. Even when referred to gynecologic oncology, patients from historically-marginalized groups have twice as long duration from diagnosis to seeing gynecologic oncology. In this project, the investigators will pilot a clinician nudge to gynecologic oncology referral and compare the impact to historical controls.

DETAILED DESCRIPTION:
The study consists of one intervention, a clinician nudge to gynecologic oncology referral. Referral to gynecologic oncology is recommended when patients are diagnosed with a complex adnexal mass on imaging (i.e., Ovarian-Adnexal Reporting and Data System [O-RADS] 4 or 5 on ultrasound or Magnetic Resonance Imaging [MRI]). When patients are identified as having a complex adnexal mass, the order will be pended by the clinical research coordinator and sent to the ordering provider with a message to sign. The message will include content about national guidelines on referral to gynecologic oncology with opt-out framed language.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 years or older
* Adnexal mass identified on imaging (i.e., O-RADS 4 or 5 on ultrasound or MRI, Codex 4 or 5 on CT scan) ordered by Penn Medicine clinician

Exclusion Criteria:

* Known diagnosis of ovarian cancer
* Patient already established in gynecologic oncology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 20 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Adoption | 30 days
  The primary implementation outcome is adoption, operationalized as the proportion of patients who are referred to gynecologic oncology within 30 days of diagnosis by study arm, to be evaluated overall and for historically marginalized patients.

SECONDARY OUTCOMES:
Gyn Onc Visits | 90 days
  The proportion of patients completing gynecologic oncology visits for surgical evaluation.
Gyn Onc Visits | 90 days
  Time to first gynecologic oncology visit (in days from radiologic or pathologic diagnosis), also to be evaluated overall and for historically marginalized patients.
Adherence to Treatment | 365 days
  Adherence to evidence-based treatment within 365 days of patient follow-up.
Progression Free and Overall Survival | 365 days
  Progression-free and overall survival within 365 days of patient follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States